CLINICAL TRIAL: NCT02609633
Title: Accu-Chek® CONNECT at School (CATS) Pediatric Study
Acronym: CATS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RD002489
Record Dates: First submitted 2015-11-18; First posted 2015-11-20 (Estimated); Results first posted 2018-05-18 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-04

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control: Usual Care - Current Diabetes Management System (DMS) (Active Comparator): Participants will perform self-monitoring of blood glucose (SMBG) for 6 months using the current DMS device. Follow-up office visits will be scheduled at Months 3 and 6 to review and discuss SMBG data and modify the type 1 diabetes (T1D) regimen as needed.
  Interventions: Device: DMS
- Interventional: Accu-Chek® CONNECT DMS (Experimental): Participants will receive training on Day 1 with the Accu-Chek® CONNECT DMS and will thereafter perform SMBG for 6 months. Follow-up office visits will be scheduled at Months 3 and 6 to review and discuss SMBG data and modify the T1D regimen as needed.
  Interventions: Device: Accu-Chek® CONNECT DMS

INTERVENTIONS:
Device: Accu-Chek® CONNECT DMS — SMBG will be performed during the 6-month study using the Accu-Chek® Aviva CONNECT monitoring device, and corresponding Smartphone app and online tracking tool.
  Arms: Interventional: Accu-Chek® CONNECT DMS
Device: DMS — SMBG will be performed during the 6-month study according to usual care, using the participant's current DMS (other than Accu-Chek® CONNECT DMS).
  Arms: Control: Usual Care - Current Diabetes Management System (DMS)

SUMMARY:
This interventional, 6-month post-marketing study is designed to evaluate the change in diabetes-related distress among parents/caregivers of school-age children and adolescents with type 1 diabetes (T1D) who are receiving multiple daily injections (MDI) therapy. Investigational sites will be assigned using cluster randomization, with approximately 10 to 20 children at each site. In order to maintain a true control group for comparison, the investigational sites will be randomly assigned to the Accu-Chek® CONNECT Diabetes Management System (DMS) or usual care/continued use of current DMS devices.

ELIGIBILITY:
Inclusion Criteria:

* Children or adolescents, aged 6 to 18 years
* Diagnosis of T1D for at least 3 months
* Currently managed with insulin Multiple Daily Injection (MDI) therapy
* Attending full-day school schedule in Grade K through 12
* Able to provide SMBG data minimum of one month prior to study start
* Currently using a compatible Smartphone with ability to download the Accu-Chek® CONNECT System App accordingly OR ability to utilize Smartphone and Accu-Chek® CONNECT System App as provided for use in study
* Adolescents (18 years) with diabetes provide written informed consent
* Children 7 to 17 years to provide age-appropriate child assent
* Parent/caregiver currently using a compatible Smartphone with ability to receive Short Message Service/Multimedia Messaging Service (SMS/MMS) messages
* Able to read/write in English and comply with study procedures, including provision of self-monitoring blood glucose (SMBG) data at least 1 month prior to the study

Exclusion Criteria:

* Current or planned use of continuous subcutaneous insulin infusions during the study period
* Use of continuous glucose monitoring or a remote data-sharing system/device (i.e. NightScout, DexCom Share, Medtronic Connect) during the study
* Pregnancy
* Clinically significant medical condition(s) such as anemia, major organ system disease, infection, psychosis, or cognitive impairment
* Requirement for chronic steroids, immunomodulatory medication, or chemotherapy in adrenal suppressive doses
* Visual impairment preventing use of the Accu-Chek® CONNECT system
* Parent/caregiver is an investigator, general practitioner, practice staff, pharmacist, research assistant, or other staff or relative of those directly involved in the study

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 196 (Actual)
Dates: Start 2015-12-28 (Actual); Primary Completion 2017-01-20 (Actual); Study Completion 2017-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lena Borsa, Study Director — Roche Diabetes Care
Locations (13):
- United States (13):
  - Pediatric Endocrinology of Phoenix, Phoenix, Arizona
  - Center of Excellence in Diabetes and Endocrinology, Sacramento, California
  - Barbara Davis Center for Childhood Diabetes, Aurora, Colorado
  - Nemours Childrens Hospital, Pensacola, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - University of South Florida College of Medicine, Tampa, Florida
  - Pediatric Endocrine Associates, Atlanta, Georgia
  - Rocky Mountain Diabetes & Osteoporosis Center, Idaho Falls, Idaho
  - Advocate Center for Pediatric Research, Oak Lawn, Illinois
  - Indiana University Riley, Carmel, Indiana
  - Childrens Hospital and Clinics of Minnesota, Saint Paul, Minnesota
  - Women and Children's Hospital of Buffalo, Buffalo, New York
  - East Caroline University - Pediatric specialty Care, Greenville, North Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Families of participants were identified and recruited from the investigators' established participant populations or from the participant populations of other physicians within the group practice, using protocol-specified inclusion and exclusion criteria.
Pre-assignment Details: Although a total of 196 parents and children/adolescents were enrolled, only the 98 children/adolescents were considered participants in the study. Baseline and adverse events data were only collected for children/adolescents.
Groups:
- Control: Usual Care - Current Diabetes Management System (DMS): Participants of enrolled families continued to use their self-monitoring of blood glucose (SMBG) for 6 months using the current DMS device.
- Interventional: Accu-Chek® CONNECT DMS: Participants of enrolled families who used Accu-Chek® CONNECT DMS for 6 months.
Period: Overall Study
Arm/Group | Control: Usual Care - Current Diabetes Management System (DMS) | Interventional: Accu-Chek® CONNECT DMS
Started | 42 | 56
Full Analysis Set (FAS) | 32 | 46
Completed | 37 | 54
Not Completed | 5 | 2
Not completed — Consent Withdrawn | 0 | 1
Not completed — Protocol Deviation | 1 | 0
Not completed — Non-Compliant with Study Procedures | 2 | 0
Not completed — Reason not Specified | 2 | 1

BASELINE CHARACTERISTICS:
Population: FAS included all eligible families that have signed an informed consent and completed (with the acceptable level of missing questions to calculate a total score) all questions on the Problem Areas in Diabetes (PAID) Parent [Parents of Youth (YP) or Parents of Teens (TP)] Questionnaire at both baseline and Visit 4 (Month 6).
Groups:
- Total: Total of all reporting groups
Arm/Group | Control: Usual Care - Current Diabetes Management System (DMS) | Interventional: Accu-Chek® CONNECT DMS | Total
Number analyzed (Participants) | 32 | 46 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.3 (3.06) | 12.6 (3.03) | 12.9 (3.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 24 | 37
  Male | 19 | 22 | 41
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black or African American | 6 | 5 | 11
  Race: White | 24 | 34 | 58
  Race: Asian | 0 | 1 | 1
  Race: Native Hawaiian or other Pacific Islander | 0 | 1 | 1
  Race: Other | 2 | 5 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic/latino:Yes | 2 | 4 | 6
  Ethnicity: Hispanic/latino:No | 30 | 42 | 72
Diabetes-Related Distress According to the PAID Child and Teen (C&T) Parent Questionnaire Score [Mean (Standard Deviation); unit: Score on a Scale] — The PAID Questionnaire encompassed 26 items. Score for each question ranges from 1-2 = "Not a Problem" to 5-6 = "Big Problem" (Child version) or 1-2 = "Not a Problem" to 5-6 = "Serious Problem" (Teen or Parent versions). The derived total score (26 questions) ranges between 26 and 156, where higher score indicates worsened condition.
  Score on a Scale | 66.2 (21.72) | 71.1 (24.53) | 69.1 (23.40)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Diabetes-Related Distress Among Parents/Caregivers According to the Problem Areas in Diabetes (PAID) Child and Teen (C&T) Parent Questionnaire Score at Month 6
Description: The PAID Questionnaire encompassed 26 items. Score for each question ranges from 1-2 = "Not a Problem" to 5-6 = "Big Problem" (Child version) or 1-2 = "Not a Problem" to 5-6 = "Serious Problem" (Teen or Parent versions). The derived total score (26 questions) ranges between 26 and 156, where higher score indicates worsened condition.
Time Frame: Baseline, Month 6
Population: The FAS included all eligible families that have signed an informed consent and completed (with the acceptable level of missing questions to calculate a total score) all questions on the PAID Parent (YP or TP) Questionnaire at both baseline and Visit 4.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control: Usual Care - Current Diabetes Management System (DMS) | Interventional: Accu-Chek® CONNECT DMS
Number analyzed (Participants) | 32 | 46
score on a scale | -0.3 (17.82) | -5.0 (21.42)

2. Secondary Outcome: Change From Baseline in Diabetes-Related Distress Among Parents/Caregivers According to the PAID C&T Child Questionnaire Score at Month 3
Description: as for outcome 1
Time Frame: Baseline, Month 3
Population: The FAS included all eligible families that have signed an informed consent and completed (with the acceptable level of missing questions to calculate a total score) all questions on the PAID Parent (YP or TP) Questionnaire at both baseline and Visit 4. Here, 'Number analysed' is the participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control: Usual Care - Current Diabetes Management System (DMS) | Interventional: Accu-Chek® CONNECT DMS
Number analyzed (Participants) | 32 | 46
score on a scale
  Baseline: number analyzed (Participants) | 31 | 43
  Baseline | 65.3 (21.42) | 70.4 (24.14)
  Change at Month 3: number analyzed (Participants) | 31 | 43
  Change at Month 3 | 4.7 (18.06) | -1.3 (19.14)

3. Secondary Outcome: Change From Baseline in Diabetes-Related Distress Among School-age Children/Adolescents and Adolescents According to the PAID C&T Child Questionnaire Score at Month 3 and 6
Description: as for outcome 1
Time Frame: Baseline, Months 3 and 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control: Usual Care - Current Diabetes Management System (DMS) | Interventional: Accu-Chek® CONNECT DMS
Number analyzed (Participants) | 32 | 46
score on a scale
  Baseline: number analyzed (Participants) | 28 | 41
  Baseline | 53.1 (26.85) | 62.2 (24.44)
  Change at Months 3: number analyzed (Participants) | 28 | 41
  Change at Months 3 | -3.0 (16.89) | 1.2 (17.44)
  Change at Months 6: number analyzed (Participants) | 28 | 39
  Change at Months 6 | -2.1 (18.00) | -0.2 (17.98)

4. Secondary Outcome: Change From Baseline in Perceived Family Conflict Among School-Age Children With Diabetes and Parent/Caregiver According to Diabetes Family Conflict Scale (DFCS) Parent Questionnaire Score at Months 3 and 6
Description: The DFCS Questionnaire has 19 questions, each question ranges in response values between 1 ("Almost Never") and 3 ("Almost Always"). The derived total score (19 questions) ranges between 19 and 57, where higher score indicates worsened condition. This questionnaire was answered by Children/adolescents and Parents.
Time Frame: Baseline, Months 3 and 6
Population: The FAS included all eligible families that have signed an informed consent and completed (with the acceptable level of missing questions to calculate a total score) all questions on the PAID Parent (YP or TP) Questionnaire at both baseline and Visit 4. The number analysed is the participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control: Usual Care - Current Diabetes Management System (DMS) | Interventional: Accu-Chek® CONNECT DMS
Number analyzed (Participants) | 32 | 46
score on a scale
  Children/adolescents DFCS Score at Baseline: number analyzed (Participants) | 30 | 41
  Children/adolescents DFCS Score at Baseline | 28.3 (10.54) | 30.3 (9.57)
  Children/adolescents DFCS Change Score at Month 3: number analyzed (Participants) | 30 | 41
  Children/adolescents DFCS Change Score at Month 3 | 0.5 (11.23) | -0.5 (9.37)
  Children/adolescents DFCS Change Score at Month 6: number analyzed (Participants) | 30 | 41
  Children/adolescents DFCS Change Score at Month 6 | -0.8 (12.09) | -0.9 (7.93)
  Parent/Caregiver DFCS Score at Baseline: number analyzed (Participants) | 29 | 41
  Parent/Caregiver DFCS Score at Baseline | 27.9 (9.13) | 27.6 (8.37)
  Parent/Caregiver DFCS Change Score at Month 3: number analyzed (Participants) | 29 | 41
  Parent/Caregiver DFCS Change Score at Month 3 | -1.6 (8.02) | -1.3 (6.15)
  Parent/Caregiver DFCS Change Score at Month 6: number analyzed (Participants) | 32 | 42
  Parent/Caregiver DFCS Change Score at Month 6 | -0.2 (7.93) | -1.6 (9.73)

5. Secondary Outcome: Change From Baseline in Affect Towards Blood Glucose Monitoring Among School-Age Children With Diabetes and Parent/Caregiver According to Blood Glucose Monitoring Communication (BGMC) Parent Questionnaire Score at Months 3 and 6
Description: The BGMC Questionnaire has 8 questions, each question ranges in response values from 1 ("Almost Never") to 3 ("Almost Always"). The derived total score ranges between 8 and 24, where higher score indicates worsened condition.
Time Frame: Baseline, Months 3 and 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control: Usual Care - Current Diabetes Management System (DMS) | Interventional: Accu-Chek® CONNECT DMS
Number analyzed (Participants) | 32 | 46
score on a scale
  Children/Adolescents BGMC Score at Baseline: number analyzed (Participants) | 29 | 43
  Children/Adolescents BGMC Score at Baseline | 12.4 (4.01) | 13.7 (3.85)
  Children/Adolescents BGMC Change Score at Month 3: number analyzed (Participants) | 29 | 43
  Children/Adolescents BGMC Change Score at Month 3 | -0.9 (2.86) | -0.1 (3.01)
  Children/Adolescents BGMC Change Score at Month 6: number analyzed (Participants) | 29 | 41
  Children/Adolescents BGMC Change Score at Month 6 | -0.4 (4.09) | -0.4 (2.90)
  Parents/Caregivers BGMC Score at Baseline: number analyzed (Participants) | 30 | 42
  Parents/Caregivers BGMC Score at Baseline | 14.4 (3.45) | 14.0 (4.03)
  Parents/Caregivers BGMC Change Score at Month 3: number analyzed (Participants) | 30 | 42
  Parents/Caregivers BGMC Change Score at Month 3 | 0.3 (2.38) | -0.7 (3.53)
  Parents/Caregivers BGMC Score Change at Month 6: number analyzed (Participants) | 31 | 41
  Parents/Caregivers BGMC Score Change at Month 6 | -0.5 (2.80) | -0.3 (4.39)

6. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin A1c (HbA1c) Among School-Age Children With Diabetes at Months 3 and 6
Description: Assessment of HbA1c is an indicator of long-term control of diabetes.
Time Frame: Baseline, Months 3 and 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Arm/Group | Control: Usual Care - Current Diabetes Management System (DMS) | Interventional: Accu-Chek® CONNECT DMS
Number analyzed (Participants) | 32 | 46
percentage of glycated hemoglobin
  Baseline: number analyzed (Participants) | 32 | 41
  Baseline | 9.3 (1.81) | 9.1 (1.80)
  Change at Month 3: number analyzed (Participants) | 32 | 41
  Change at Month 3 | -0.1 (0.94) | -0.1 (1.25)
  Change at Month 6: number analyzed (Participants) | 32 | 39
  Change at Month 6 | -0.1 (1.10) | -0.1 (1.44)

7. Secondary Outcome: Change From Baseline in Percentage of Blood Glucose (BG) Measurements Among School-Age Children With Diabetes at Months 3 and 6 Within Glucose Target Range
Description: The percentage of target range measurements was defined as the number of within target range readings in the interval divided by the total number of BG checks in the interval.
Time Frame: Baseline, Months 3 and 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of blood glucose measurements
Arm/Group | Control: Usual Care - Current Diabetes Management System (DMS) | Interventional: Accu-Chek® CONNECT DMS
Number analyzed (Participants) | 32 | 46
percentage of blood glucose measurements
  Target Range 70-160 mg/dl: Baseline: number analyzed (Participants) | 30 | 38
  Target Range 70-160 mg/dl: Baseline | 39.0 (18.91) | 30.0 (19.42)
  Target Range 70-160 mg/dl: Change at Month 3: number analyzed (Participants) | 30 | 38
  Target Range 70-160 mg/dl: Change at Month 3 | -3.9 (25.56) | 2.8 (12.46)
  Target Range 70-160 mg/dl: Change at Month 6: number analyzed (Participants) | 30 | 37
  Target Range 70-160 mg/dl: Change at Month 6 | -4.8 (22.13) | 0.5 (15.60)
  Target Range 80-180 mg/dl: Baseline: number analyzed (Participants) | 30 | 38
  Target Range 80-180 mg/dl: Baseline | 41.4 (19.03) | 31.9 (20.26)
  Target Range 80-180 mg/dl: Change at Month 3: number analyzed (Participants) | 30 | 38
  Target Range 80-180 mg/dl: Change at Month 3 | -4.6 (25.60) | 3.8 (12.99)
  Target Range 80-180 mg/dl: Change at Month 6: number analyzed (Participants) | 30 | 37
  Target Range 80-180 mg/dl: Change at Month 6 | -4.2 (22.68) | 1.4 (14.96)

8. Secondary Outcome: Change From Baseline Blood Glucose Variability Among School-Age Children With Diabetes at Months 3 and 6
Description: Glycemic variability, expressed as mean of all blood glucose(BG) readings per subject within the interval. BG variability was defined as standard deviation (SD) of all glucose readings over the interval.
Time Frame: Baseline, Months 3 and 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dl)
Arm/Group | Control: Usual Care - Current Diabetes Management System (DMS) | Interventional: Accu-Chek® CONNECT DMS
Number analyzed (Participants) | 32 | 46
milligrams per deciliter (mg/dl)
  Baseline: number analyzed (Participants) | 30 | 38
  Baseline | 94.0 (30.84) | 99.2 (32.38)
  Change at Month 3: number analyzed (Participants) | 30 | 38
  Change at Month 3 | -1.3 (30.47) | -2.3 (21.78)
  Change at Month 6: number analyzed (Participants) | 30 | 37
  Change at Month 6 | 2.8 (20.39) | -3.4 (23.48)

9. Secondary Outcome: Change From Baseline in Percentage of Hypoglycemic BG Measurements Among School-Age Children With Diabetes at Months 3 and 6
Description: A measurement was defined as hypoglycemic if the glucose value was below 70 mg/dl or below 60 mg/dl or below 50 mg/dl.
Time Frame: Baseline, Months 3 and 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of hypoglycemic measurements
Arm/Group | Control: Usual Care - Current Diabetes Management System (DMS) | Interventional: Accu-Chek® CONNECT DMS
Number analyzed (Participants) | 32 | 46
percentage of hypoglycemic measurements
  Hypoglycemia (< 70 mg/dl): Baseline: number analyzed (Participants) | 30 | 38
  Hypoglycemia (< 70 mg/dl): Baseline | 4.4 (6.20) | 5.4 (6.64)
  Hypoglycemia (< 70 mg/dl) Change at Months 3: number analyzed (Participants) | 30 | 38
  Hypoglycemia (< 70 mg/dl) Change at Months 3 | 1.7 (7.07) | 0.1 (7.55)
  Hypoglycemia (< 70 mg/dl): Change at Months 6: number analyzed (Participants) | 30 | 37
  Hypoglycemia (< 70 mg/dl): Change at Months 6 | 1.3 (6.22) | 1.6 (9.04)
  Hypoglycemia (< 60 mg/dl): Baseline: number analyzed (Participants) | 30 | 38
  Hypoglycemia (< 60 mg/dl): Baseline | 2.2 (4.28) | 2.8 (4.64)
  Hypoglycemia (< 60 mg/dl): Change at Month 3: number analyzed (Participants) | 30 | 38
  Hypoglycemia (< 60 mg/dl): Change at Month 3 | 0.8 (5.03) | -0.0 (5.53)
  Hypoglycemia (< 60 mg/dl): Change at Month 6: number analyzed (Participants) | 30 | 37
  Hypoglycemia (< 60 mg/dl): Change at Month 6 | 0.5 (5.10) | 0.1 (6.37)
  Hypoglycemia (< 50 mg/dl): Baseline: number analyzed (Participants) | 30 | 38
  Hypoglycemia (< 50 mg/dl): Baseline | 1.0 (2.76) | 1.4 (3.45)
  Hypoglycemia (< 50 mg/dl): Change at Month 3: number analyzed (Participants) | 30 | 38
  Hypoglycemia (< 50 mg/dl): Change at Month 3 | -0.4 (3.08) | -0.5 (3.74)
  Hypoglycemia (< 50 mg/dl): Change at Month 6: number analyzed (Participants) | 30 | 37
  Hypoglycemia (< 50 mg/dl): Change at Month 6 | 0.1 (3.21) | -0.6 (3.98)

10. Secondary Outcome: Percentage of Participants Who Frequently Used Accu-Chek® CONNECT Diabetes Management System According to a Questionnaire About Usability
Description: Percentage of participants who frequently used Accu-Chek® CONNECT Diabetes Management System (blood sugar meter [BSM], phone application [PA] and web portal [WP]) according to the questionnaire about usability answered by children/adolescents and Parent were reported. Here, in parent post questionnaire for usability the sum of percentages are not equal to 100%, because percentage is based on n=44.
Time Frame: Month 6
Population: The FAS included all eligible families that have signed an informed consent and completed (with the acceptable level of missing questions to calculate a total score) all questions on the PAID Parent (YP or TP) Questionnaire at both baseline and Visit 4. Here, 'Number analyzed' is the participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Interventional: Accu-Chek® CONNECT DMS
Number analyzed (Participants) | 46
percentage of participants
  Children/Adolescents: BSM - Frequently Used: number analyzed (Participants) | 41
  Children/Adolescents: BSM - Frequently Used | 97.6
  Children/Adolescents: BSM - Frequently Not Used: number analyzed (Participants) | 41
  Children/Adolescents: BSM - Frequently Not Used | 2.4
  Children/Adolescents: PA - Frequently Used: number analyzed (Participants) | 41
  Children/Adolescents: PA - Frequently Used | 78.0
  Children/Adolescents: PA - Frequently Not Used: number analyzed (Participants) | 41
  Children/Adolescents: PA - Frequently Not Used | 22.0
  Children/Adolescents: WP - Frequently Used: number analyzed (Participants) | 41
  Children/Adolescents: WP - Frequently Used | 36.6
  Children/Adolescents: WP - Frequently Not Used: number analyzed (Participants) | 41
  Children/Adolescents: WP - Frequently Not Used | 63.4
  Parents: BSM - Frequently Used: number analyzed (Participants) | 44
  Parents: BSM - Frequently Used | 86.4
  Parents: BSM - Frequently Not Used: number analyzed (Participants) | 44
  Parents: BSM - Frequently Not Used | 13.6
  Parents: PA - Frequently Used: number analyzed (Participants) | 43
  Parents: PA - Frequently Used | 79.5
  Parents: PA - Frequently Not Used: number analyzed (Participants) | 43
  Parents: PA - Frequently Not Used | 18.2
  Parents: WP - Frequently Used: number analyzed (Participants) | 40
  Parents: WP - Frequently Used | 47.7
  Parents: WP - Frequently Not Used: number analyzed (Participants) | 40
  Parents: WP - Frequently Not Used | 43.2

11. Secondary Outcome: Percentage of Participants With Participants Preference for Accu-Chek® CONNECT Diabetes Management System With Previous Technology/Process
Description: Participants preference the Accu-Chek® CONNECT process compared with previous technology/process assessed by questionnaire including following questions; Q 1: Felt more sure of myself using the system, Q 2: Less worried about low BG than used to be, Q 3: Would rather use the system than what used before, Q 4: Felt safer managing diabetes using system than what used before, Q 5: Friends with diabetes should also use the system. Questionnaire was answered by children/adolescents and parents. Here, in children/adolescents post questionnaire for preference the percentage sum is not equal to 100%, because percentage is based on n=41.
Time Frame: Month 6
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Interventional: Accu-Chek® CONNECT DMS
Number analyzed (Participants) | 46
percentage of participants
  Children/Adolescents: Q 1- Mostly Agree: number analyzed (Participants) | 40
  Children/Adolescents: Q 1- Mostly Agree | 90.2
  Children/Adolescents: Q 1- Mostly Disagree: number analyzed (Participants) | 40
  Children/Adolescents: Q 1- Mostly Disagree | 7.3
  Children/Adolescents: Q 2- Mostly Agree: number analyzed (Participants) | 41
  Children/Adolescents: Q 2- Mostly Agree | 90.2
  Children/Adolescents: Q 2- Mostly Disagree: number analyzed (Participants) | 41
  Children/Adolescents: Q 2- Mostly Disagree | 9.8
  Children/Adolescents: Q 3- Mostly Agree: number analyzed (Participants) | 41
  Children/Adolescents: Q 3- Mostly Agree | 90.2
  Children/Adolescents: Q 3- Mostly Disagree: number analyzed (Participants) | 41
  Children/Adolescents: Q 3- Mostly Disagree | 9.8
  Children/Adolescents: Q 4- Mostly Agree: number analyzed (Participants) | 41
  Children/Adolescents: Q 4- Mostly Agree | 90.2
  Children/Adolescents: Q 4- Mostly Disagree: number analyzed (Participants) | 41
  Children/Adolescents: Q 4- Mostly Disagree | 9.8
  Children/Adolescents: Q 5- Mostly Agree: number analyzed (Participants) | 41
  Children/Adolescents: Q 5- Mostly Agree | 85.4
  Children/Adolescents: Q 5- Mostly Disagree: number analyzed (Participants) | 41
  Children/Adolescents: Q 5- Mostly Disagree | 14.6
  Parent: Q 1- Mostly Agree: number analyzed (Participants) | 44
  Parent: Q 1- Mostly Agree | 90.9
  Parent: Q 1- Mostly Disagree: number analyzed (Participants) | 44
  Parent: Q 1- Mostly Disagree | 9.1
  Parent: Q 2- Mostly Agree: number analyzed (Participants) | 44
  Parent: Q 2- Mostly Agree | 88.6
  Parent: Q 2- Mostly Disagree: number analyzed (Participants) | 44
  Parent: Q 2- Mostly Disagree | 11.4
  Parent: Q 3- Mostly Agree: number analyzed (Participants) | 44
  Parent: Q 3- Mostly Agree | 90.9
  Parent: Q 3- Mostly Disagree: number analyzed (Participants) | 44
  Parent: Q 3- Mostly Disagree | 9.1
  Parent: Q 4- Mostly Agree: number analyzed (Participants) | 44
  Parent: Q 4- Mostly Agree | 90.9
  Parent: Q 4- Mostly Disagree: number analyzed (Participants) | 44
  Parent: Q 4- Mostly Disagree | 9.1
  Parent: Q 5- Mostly Agree: number analyzed (Participants) | 44
  Parent: Q 5- Mostly Agree | 95.5
  Parent: Q 5- Mostly Disagree: number analyzed (Participants) | 44
  Parent: Q 5- Mostly Disagree | 4.5

12. Secondary Outcome: Percentage of Participants With Overall Treatment Satisfaction With the Use of Accu-Chek® CONNECT Diabetes Management System According to a Questionnaire
Description: Percentage of participants with overall treatment satisfaction with the use of Accu-Chek® CONNECT Diabetes Management system according to the questionnaire answered by children/adolescents and parents were reported.
Time Frame: Month 6
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Interventional: Accu-Chek® CONNECT DMS
Number analyzed (Participants) | 46
percentage of participants
  Children/adolescents: Satisfied: number analyzed (Participants) | 40
  Children/adolescents: Satisfied | 87.8
  Children/adolescents: Not Satisfied: number analyzed (Participants) | 41
  Children/adolescents: Not Satisfied | 9.8
  Parent: Satisfied: number analyzed (Participants) | 41
  Parent: Satisfied | 88.4
  Parent: Not Satisfied: number analyzed (Participants) | 41
  Parent: Not Satisfied | 4.7

ADVERSE EVENTS:
Time Frame: Baseline up to Month 6
Description: The Safety Population included all participants.
Arm/Group | Control: Usual Care - Current Diabetes Management System (DMS) | Interventional: Accu-Chek® CONNECT DMS
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/56
Serious Adverse Events (participants affected / at risk) | 4/42 | 2/56
Other Adverse Events (participants affected / at risk) | 28/42 | 6/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control: Usual Care - Current Diabetes Management System (DMS) (N=42) | Interventional: Accu-Chek® CONNECT DMS (N=56)
Vomiting (Gastrointestinal disorders) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 2 | 0
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Control: Usual Care - Current Diabetes Management System (DMS) (N=42) | Interventional: Accu-Chek® CONNECT DMS (N=56)
Gastroenteritis viral (Infections and infestations) | 4 | 0
Upper respiratory tract infection (Infections and infestations) | 5 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 27 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2015-08-27): https://cdn.clinicaltrials.gov/large-docs/33/NCT02609633/Prot_000.pdf
  • Statistical Analysis Plan (2016-06-27): https://cdn.clinicaltrials.gov/large-docs/33/NCT02609633/SAP_001.pdf